CLINICAL TRIAL: NCT04525963
Title: The Effect of Operating Room Nurse Visit Prior to Cardiac Surgery on Patients's Anxiety, Pain and Analgesic Use
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nurgül Arpag (Other)
Responsible Party: Sponsor-Investigator, Nurgül Arpag, Lecturer, Istanbul University - Cerrahpasa
Organization: Istanbul University - Cerrahpasa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NArpag
Record Dates: First submitted 2020-08-17; First posted 2020-08-25 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Postoperative Anxiety; Pain; Postoperative Pain Management
Keywords: Anxiety; Surgical anxiety; Surgical pain; Open heart surgey; Nursing
MeSH Terms: conditions — Pain; Anxiety Disorders | interventions — Patient Education as Topic

STUDY DESIGN:
Intervention Model Description: A quasi-experimental pre-test post-test control group design in non-randomized groups study,to determine the effect of the preoperative visit by the operating room nurse on the postoperative anxiety level and pain severity of patients undergoing open heart surgery
Who Masked: Outcomes Assessor
Masking Description: Single blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Intervention Arm (Experimental): :In the experimental group,the operating room nurse, who is given intervention training , will be provided to visit the patient before surgery. After the verbal training of the operating room nurse, a printed booklet will be left for the patient to read.
  Assigned Interventions The level of anxiety experienced by the patients increases the postoperative perception and analgesic need, increasing the sequence and anesthetic substance. For these reasons, there is a need for studies to reduce pain distribution and severity by directly dealing with pre- and postoperative anxiety and anxiety levels. Similarly, the role of the operating room nurse in reducing patient anxiety is increasingly recognized. It is observed that the pre-operative visit and education reduce the pre-operative anxiety level in patients undergoing surgical intervention, and the pre-operative visit of the operating room nurse is on the agenda.
  Interventions: Other: Preoperative visit of the operating room nurse and patient education
- No Intervention (No Intervention): There will be no intervention in the control group. The procedures of the institution will be applied before and after the operation.

INTERVENTIONS:
Other: Preoperative visit of the operating room nurse and patient education — The operating room nurse, who is given intervention training, will visit the patient before the operation. After the oral training of the operating room nurse, a printed booklet will be left for the patient to read.
  Arms: Experimental: Intervention Arm

SUMMARY:
This study was planned as a quasi-experimental pre-test post-test control group design in non-randomized groups to determine the effect of the preoperative visit by the operating room nurse on the postoperative anxiety level and pain severity of patients undergoing open heart surgery.After approval of the ethics committee and institutional permission, 64 patients who were operated in Cardiovascular Surgery between September 1, 2020 and April 1, 2020 and met the inclusion criteria will be included in the study.Sample size and power analysis of the research was calculated by using the Clinical Calculator program,reported academic studies was determined as effect value (size) d = 2.0935, α = 0.05 (margin of error), 1-β = 0.80 (Power).It was decided to include 64 people (32 per group). operated with the CPB (cardiopulmonary bypass) method were included. The assignment to the control group and the experimental group of patients who meet the inclusion criteria and agree to participate in the study will be made with the random numbers table created using the create number function in the Excel program.

DETAILED DESCRIPTION:
Patients who will undergo cardiac surgery between 01 September 2020 and 01 April 2021 and meet the inclusion criteria will be able to participate in the study with their verbal and written consents. The assignment of the patients to the control or experimental group will be done with the random numbers table created using the generate number function in the Excel program. This study will be conducted in 64 patients (32 patients in each group) who will be operated in cardiac surgery at Istanbul Yeni Yüzyıl University GOP hospital. In order to determine the postoperative anxiety and pain management effects of the patient visit of the operating room nurse, the pre-test-post-test control group design will be made quasi-experimental in non-randomized groups. The variables of the study were anxiety, pain, and analgesic use. As data collection tools, 'Sampling Criteria Form' will be used for sampling and 'State Trait Anxiety Scale I-II ' will be used for anxiety assessment. "VAS (Visual Analogue Scale)" will be used for pain assessment, and "Analgesic Follow-up Form" developed by the researcher will be used for the recording of analgesics. The "Data Recording Form" created by the researcher will be used to record the demographic and medical data of the patients.

The researcher will apply the "State-Trait Anxiety Scale" to determine the level of anxiety after visiting the patient's room and obtaining verbal and written permission from the patient. If the patient is in the control group, it will be ensured that the institutional procedures are implemented and followed without any intervention (without visiting and verbal training printed booklet). In the experimental group,the operating room nurse, who is given intervention training , will be provided to visit the patient before surgery. After the verbal training of the operating room nurse, a printed booklet will be left for the patient to read. It will be ensured that the nurse visiting the patient in her room will be welcomed in the operating room. After the operation, the pain level of the patient will be monitored by the Visual Assessment Scale (VAS) in the intensive care and inpatient floor. Pain level and use of analgesics will be monitored at the first 72 hours and thereafter until the thoracic tubes are removed. The analgesics ordered for the patient will be recorded according to time, name, dose and route of administration. For these records, "Analgesic Registration Form" developed by the researcher will be used.Patients with prolonged intensive care stay (over 96 hours) and returning to intensive care will be excluded from the evaluation. If these patients are excluded from the study, an "intention to treat" (ITT) analysis will be performed to assess the realistic effect of the intervention. "State-Trait Anxiety Scale" will be applied again by the researcher on the 24th hour to determine the postoperative anxiety level of all patients.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-75,
* Having surgery with a cardiopulmonary bypass (CPB)
* no psychiatric diagnosis and drug use
* first cardiovascular experience
* having elective and planned surgery
* being literate and speaking Turkish
* Patients who agree to participate in the study will be included in the study.

Exclusion Criteria:

* Emergency surgery,
* Being under the age of 18
* psychiatric diagnosis and drug use
* Not using cardiopulmonary bypass
* have previously had open heart surgery
* be illiterate
* not understanding and speaking Turkish
* staying in intensive care for more than 96 hours or returning to intensive care
* refuse to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2021-02-20 (Estimated); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
1. Anxiety before and after surgery / State Trait Anxiety Scale I-II' Score | In the preoperative period, the anxiety scale score will be evaluated within the last 18 hours. In the postoperative period, the anxiety scale score will be evaluated within the first 18 hours.
  Anxiety severity will be assessment with 'State Trait Anxiety Scale I-II' State anxiety scale-I,it involves the marking of (1) none, (2) a little, (3) quite, (4) completely one of the options of the individual at a given moment according to the current emotions of the items of the scale.
  The trait anxiety scale-II, requires one out of four options to mark how the individual usually feels (1) almost never, (2) sometimes, (3) much time, (4) almost always.
  There are two types of expressions in the scales, are called direct or inverted expressions. Direct expressions, negative emotions; reversed expressions express positive feelings.
2. Postoperative pain severity | In the postoperative period, the severity of the pain is evaluated until the end of the first 24 hours.
  Pain severity assessment with Visual Assessment Scale (VAS) Score: 0-10; 0- No Pain, 10- Worst pain
3. Measurement of postoperative analgesic use | The analgesics used in the postoperative period are evaluated until the end of the first 24 hours.
  Monitoring analgesic use:time, name, type, dose, frequency and route of administration will be tracked with the Analgesic Registration form.

CONTACTS AND LOCATIONS:
Overall Officials: Denyan Mansuroğlu, Prof., Principal Investigator — Istanbul Yeni Yüzyıl University GOP Hospital; Deniz S Öztekin, Prof., Study Director — Istanbul University - Cerrahpasa; Nurgül Arpag, MSC, Study Chair — Istanbul University - Cerrahpasa

IPD SHARING:
Plan to Share IPD: No